CLINICAL TRIAL: NCT03290885
Title: Combined Use of Contact Aspiration and the Stent Retriever Technique Versus Stent Retriever Alone for Recanalisation in Acute Cerebral Infarction: the Randomized ASTER2 Study
Brief Title: Combined Use of Contact Aspiration and the Stent Retriever Technique Versus Stent Retriever Alone for Recanalisation in Acute Cerebral Infarction
Acronym: ASTER2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017014F; 2016-A01735-46 (Other: ANSM)
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined use of contact aspiration and stent retriever (Experimental): Combined use of contact aspiration and stent retriever mechanical thrombectomy for recanalization
  Interventions: Combination Product: Combined contact aspiration/Stent Retriever Technique
- Stent retriever mechanical thrombectomy alone (Active Comparator): Stent retriever mechanical thrombectomy alone for recanalisation
  Interventions: Device: Stent retriever technique

INTERVENTIONS:
Combination Product: Combined contact aspiration/Stent Retriever Technique — Combined contact aspiration/SR is performed using a balloon-guide catheter (BGC). A 0.021 to 0.027 inch inner lumen microcatheter with a 0.014 to 0.016 inch micro-wire inside is introduced into a large-bore aspiration catheter and this construct is introduced into BGC. The BGC is placed into the origin of the cervical internal carotid artery (ICA). The catheter is advanced past the thrombus over the micro-wire to allow the SR deployment. The SR is deployed across the occlusion. Then the large bore distal access catheter is advanced to contact the proximal edge of the SR. The aspiration pump is connected to the large bore distal access catheter. After at least 90 sec, the SR and the large bore distal access catheter are pulled out as an unit from the BGC and the patient. Manual aspiration is also be applied to the BGC during the pull-out manoeuver which is performed after the temporary inflation of the balloon at the tip of the BGC to ensure flow arrest into the carotid
  Arms: Combined use of contact aspiration and stent retriever
Device: Stent retriever technique — The technique used should be in accordance with the device instruction for use. A large bore balloon guide catheter has to be placed into the cervical ICA.
  A suitable delivery microcatheter is navigated over a micro-wire into the occluded major coronary artery MCA and across the occlusion. A control superselective angiogram may be used to document the extent of occlusion and thrombus. The stent retriever device is then deployed across the occlusion.
  After at least 90 seconds, removal should occur with proximal occlusion by inflation of the balloon guide catheter.
  Arms: Stent retriever mechanical thrombectomy alone

SUMMARY:
Mechanical thrombectomy (MT) with a stent retriever (SR) device is now the standard intervention in ischemic stroke with large vessel occlusion. Favorable outcome is strongly associated with the successful reperfusion status. New device of MT such as contact aspiration seems promising to increase reperfusion status and clinical outcome.

The main hypothesis is to show the superiority of combining the use of contact aspiration with a stent retriever compared to a stent retriever alone in treatment of acute stroke due to proximal arterial occlusion.

The primary endpoint is the rate of perfect reperfusion score at the end of the endovascular procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older (i.e., candidates must have had their 18th birthday)
* Groin puncture carried out within 8 hours of first symptoms
* Neuroimaging demonstrates large vessel proximal occlusion (distal ICA through MCA bifurcation, M1 or M2)
* Consenting requirements met according to French laws.
* With or without intravenous thrombolysis

Exclusion Criteria:

* Absence of large vessel occlusion on non-invasive imaging
* Known or suspected pre-existing (chronic) large vessel occlusion in the symptomatic territory
* Suspected pregnancy; if, a woman is of childbearing potential, a urine or serum beta human chorionic gonadotropin (betaHCG) test is positive.
* Severe contrast medium allergy or absolute contraindication to iodinated agents.
* Patient has severe or fatal comorbidities that will likely prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.
* Acute ischemic stroke involving posterior circulation (vertebrobasilar occlusion)
* Angiographic evidence of carotid dissection or tandem cervical occlusion or stenosis requiring treatment.
* Patients benefiting from a legal protection
* Non-membership of a national insurance scheme
* Opposition of the patient or (in case of inclusion as a matter of urgency) of the trustworthy person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Perfect reperfusion rate | 24 hours
  Perfect reperfusion rate at the end of angiography defined as a Thrombolysis In Cerebral Infarction (TICI) 2c/3 score (TICI score = Thrombolysis In Cerebral Infarction)

SECONDARY OUTCOMES:
Rate of successful reperfusion | 24 hours
  Rate of successful reperfusion (mTICI 2b/2c/3), and complete reperfusion (mTICI3) at end of endovascular procedure
Rate of perfect (mTICI 2c/3), successful reperfusion (mTICI 2b/2c/3), and complete reperfusion (mTICI3) after the frontline strategy | 24 hours
Time from groin puncture to achieve TICI 2c or better revascularization | 24 hours
  Time from groin puncture to achieve TICI 2c or better revascularization
Time between groin puncture to clot contact and clot contact to maximum reperfusion | 24 hours
  Time between groin puncture to clot contact and clot contact to maximum reperfusion
Modified Rankin scale (mRs) | 90 days
  Global disability assessed by overall distribution of mRs at 90-days
Rate of favorable functional independence | 90 days
  Rate of favorable functional independence defined as a mRS 0-2 at 90 days
Rate of excellent functional outcome | 90 days
  Rate of excellent functional outcome defined as a Modified Rankin scale (mRS) 0-1 at 90 days
NIHSS score | 24 hours
  Change in NIHSS from baseline to 24 hours (delta NIHSS)
Rate of symptomatic and asymptomatic intracerebral hemorrhage | 24 hours
  Rate of symptomatic and asymptomatic intracerebral hemorrhage at MRI 24h after thrombectomy (according the third European Cooperative Acute Stroke Study (ECASS3) classification) (independent core lab adjudication).
Rate of parenchymal hematoma | 90 days
Rate of all-cause mortality | 90 days
Rate of periprocedural complications | 90 days
  - Rate of periprocedural complications: Occurrence of emboli to new territory (ENT), vasospasm, dissection, or perforation.
Average cost per patient | 90 days
  Average cost per patient with complete recanalization

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lapergue, MD, Principal Investigator — Hôpital Foch; Michel Piotin, MD, Study Chair — Fondation Ophtalmologique de Rothschild
Locations (11):
- France (11):
  - CHU Bordeaux, Bordeaux
  - CHU Limoges, Limoges
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Fondation Ophtalmologique Rotschild, Paris
  - Kremlin-Bicêtre (APHP), Paris
  - La Pitié-Salpétrière (APHP), Paris
  - Lariboisière (APHP), Paris
  - CHU Rennes, Rennes
  - Hôpital Foch, Suresnes

REFERENCES:
- [Derived] Sgreccia A, Desilles JP, Costalat V, Dargazanli C, Bourcier R, Tessier G, Rouchaud A, Saleme S, Spelle L, Caroff J, Marnat G, Barreau X, Clarencon F, Shotar E, Eugene F, Houdart E, Gory B, Zhu F, Labreuche J, Piotin M, Lapergue B, Consoli A; ASTER2 Investigators. Combined Technique for Internal Carotid Artery Terminus or Middle Cerebral Artery Occlusions in the ASTER2 Trial. Stroke. 2024 Feb;55(2):376-384. doi: 10.1161/STROKEAHA.123.045227. Epub 2023 Dec 21. PMID 38126181
- [Derived] Lapergue B, Blanc R, Costalat V, Desal H, Saleme S, Spelle L, Marnat G, Shotar E, Eugene F, Mazighi M, Houdart E, Consoli A, Rodesch G, Bourcier R, Bracard S, Duhamel A, Ben Maacha M, Lopez D, Renaud N, Labreuche J, Gory B, Piotin M; ASTER2 Trial Investigators. Effect of Thrombectomy With Combined Contact Aspiration and Stent Retriever vs Stent Retriever Alone on Revascularization in Patients With Acute Ischemic Stroke and Large Vessel Occlusion: The ASTER2 Randomized Clinical Trial. JAMA. 2021 Sep 28;326(12):1158-1169. doi: 10.1001/jama.2021.13827. PMID 34581737